CLINICAL TRIAL: NCT07329140
Title: Outcomes of Robotic-Assisted Urological Surgery
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202510125RINB
Record Dates: First submitted 2025-12-04; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Outcome Assessment
Keywords: robotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective review of the patients who underwent urological robotic surgeries.

DETAILED DESCRIPTION:
Outcomes of the operations are reviewed.

ELIGIBILITY:
Inclusion Criteria: Patients who underwent robotic-assited urological surgery -

Exclusion Criteria: age under 18

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent robotic-assited urological surgery
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2026-11-27 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Perioperative outcomes | 1 year
  Oncological and functional outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan